CLINICAL TRIAL: NCT04082767
Title: Sedation Efficacy of Dexmedetomidine Versus Midazolam in Critically Ill Ventilated Children
Status: Unknown | Phase: Phase 3 | Type: Interventional
Last Known Status: Recruiting
Sponsor: Douglas Fraser (Other)
Responsible Party: Sponsor-Investigator, Douglas Fraser, Paediatric Intensivist, London Health Sciences Centre Research Institute OR Lawson Research Institute of St. Joseph's
Organization: London Health Sciences Centre Research Institute OR Lawson Research Institute of St. Joseph's (Other)
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Supportive Care
Other Study IDs: PEDSED01
Record Dates: First submitted 2019-08-28; First posted 2019-09-09 (Actual); Last update posted 2023-12-11 (Actual); Status verified 2023-12

CONDITIONS: Mechanically Ventilated, Critically Ill Children
Keywords: sedation, delirium, pediatric, critical care
MeSH Terms: conditions — Delirium | interventions — Dexmedetomidine; Midazolam

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Dexmedetomidine (Active Comparator)
  Interventions: Drug: Precedex
- Midazolam (Active Comparator)
  Interventions: Drug: Midazolam

INTERVENTIONS:
Drug: Precedex — Precedex, dexmedetomidine hydrochloride, IV, 4mcg/mL, infusion duration determined by the clinical care team
  Other Names: dexmedetomidine
  Arms: Dexmedetomidine
Drug: Midazolam — Midazolam, IV, 5mg/mL (for patients more than 10kg), 1mg/mL (for patients 2-10kg), infusion duration determined by the clinical care team
  Arms: Midazolam

SUMMARY:
There is a significant lack of adequately powered randomized clinical trial (RCT) data to determine the comparative safety and effectiveness of sedative treatments in pediatric patients. In many centres the standard of care for sedation in pediatric critical care unit (PCCU) patients includes the use of benzodiazepines despite the known negative effects of increased patient agitation and delirium, which can contribute to longer PCCU and hospital length of stay (LOS). The use of an alternative sedative, dexmedetomidine may reduce negative effects in this population. As such, the investigators plan to conduct a well designed comparative RCT to determine the most effective and safest sedative in this vulnerable population utilizing clinical assessments of sedation levels and delirium instance, electroencephalography (EEG) analysis and patient important outcomes.

ELIGIBILITY:
Inclusion Criteria:

1. Age is 1 month to 18 years inclusive
2. The patient is intubated and is expected to remain intubated for at least the next 48 hours
3. The patient has not been receiving mechanical ventilation for more than 72 hours
4. The patient must already be receiving an opioid infusion per PCCU Guidelines for Sedation & Analgesia for Procedures Outside O.R. and need additional sedation.

Exclusion Criteria:

1. Admission is a consequence of suspected or proven drug overdose
2. Patient is receiving dialysis
3. Known pregnancy or lactation
4. Neuromuscular blockade other than for intubation
5. General anesthesia in the 24 hours prior to study initiation
6. An acquired Central Nervous System (CNS) condition (i.e. encephalitis, traumatic brain injury) resulting in ongoing dysfunction or an acquired condition resulting in ongoing dysfunction
7. Acute hepatitis or severe liver disease
8. Known history of sensitivity to midazolam and/or dexmedetomidine or their constituents
9. Systolic blood pressure (SBP) below 5th percentile for two consecutive measurements
10. Heart rate (HR) below 5th percentile for two consecutive measurements
11. Death is deemed to be imminent or inevitable during the admission and either the intensivist or substitute decision maker is not committed to full active resuscitation
12. Previous enrollment into the study

Ages: 1 Month to 17 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 120 (Estimated)
Dates: Start 2021-06-08 (Actual); Primary Completion 2024-09 (Estimated); Study Completion 2024-09 (Estimated)

PRIMARY OUTCOMES:
Target Sedation Range | Up to 14 days post-randomization
  The percentage of time spent within target sedation range, defined as COMFORT Behaviour Scale score of 11-22, which will be assessed at minimum every 4 hours.

SECONDARY OUTCOMES:
Delirium | Up to 14 days post-randomization
  Prevalence of delirium using the Cornell Assessment of Pediatric Delirium (CAPD) tool
Delirium | Up to 14 days post-randomization
  Duration of delirium using the Cornell Assessment of Pediatric Delirium (CAPD) tool
Delirium | Up to 14 days post-randomization
  Prevalence of delirium using raw and quantitative EEG
Delirium | Up to 14 days post-randomization
  Duration of delirium using raw and quantitative EEG
Duration of mechanical ventilation | Up to 28 days post-randomization
  Mechanical ventilation-free days through day 28 will be calculated as 28 minus the duration of mechanical ventilation. Participants who die, are still receiving mechanical ventilation, or are transferred from the PCCU still receiving mechanical ventilation by day 28 will be censored at 28 days and assigned zero mechanical ventilation-free days
PCCU Length of Stay | Up to 90 days post-randomization
  Length of stay will be calculated from the time of PCCU admission to the time of PCCU discharge.
Hospital Length of Stay | Up to 90 days post-randomization
  Hospital Length of Stay will be calculated from the time of PCCU admission to the time of physical hospital discharge.
Adverse event (AE) occurrence | Randomization to 90 days post-randomization
  Documentation of treatment related adverse events including blood pressure/heart rate changes requiring decreasing or discontinuation of study drug or intervention, delirium requiring medical treatment, any unplanned extubation or line removals, aspirations, ulcerations, etc.determined to result from inadequate sedation
Quantification of sleep stages and sleep quality assessment | Up to 14 days post-randomization
  Visual and automated scoring of sleep stages from EEG recordings Stage 1 sleep: scored when more than 15 seconds of the epoch is made up of theta activity (4to7 Hz) Stage 2 sleep: predominant theta activity (4 to 7 Hz) and occasional quick bursts of faster activity Stage 3/4 sleep: marked by high-amplitude slow waves Rapid eye movement (REM) sleep: characterized by low-amplitude, mixed-frequency theta waves, intermixed with some alpha waves (usually 1 to 2 Hz slower than wake).
Pharmacokinetics - Maximum plasma concentration (Cmax) | Up to 14 days post-randomization
  Maximum plasma concentration (Cmax)
Pharmacokinetics - Area under the plasma concentration-time curve (AUC) | Up to 14 days post-randomization
  Area under the plasma concentration-time curve (AUC)
Use of open label boluses for sedation - number | Up to 14 days post-randomization
  Number of boluses (opioid and benzodiazepine) administered during the treatment period
Use of open label boluses for sedation - total dose | Up to 14 days post-randomization
  Total dose of boluses (opioid and benzodiazepine) administered during the treatment period

OTHER OUTCOMES:
Economic Analysis | Up to 90 days post-randomization
  The investigators will perform an economic evaluation during this pilot trial. This will be cost estimate analysis based on approximate costs incurred daily in the PCCU. Costs will be determined at discharge from estimated cost per day of admission to the PCCU.

CONTACTS AND LOCATIONS:
Overall Officials: Douglas D Fraser, MD., PhD, Principal Investigator — London Health Sciences Centre Research Institute OR Lawson Research Institute of St. Joseph's
Locations (1):
- Children's Hospital - London Health Sciences Centre, London, Ontario, Canada

IPD SHARING:
Plan to Share IPD: No